CLINICAL TRIAL: NCT05308862
Title: Prevention of Pressure Ulcers, Malnutrition, Poor Oral Health and Falls Among Older Persons Receiving Municipal Health Care and Are Registered in the Quality Registry Senior Alert
Brief Title: PROSENIOR. Prevention of Pressure Ulcers, Malnutrition, Poor Oral Health and Falls Among Older Persons Receiving Municipal Health Care and Are Registered in the Quality Registry Senior Alert
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Collaborators: Malmö City (Unknown)
Responsible Party: Principal Investigator, Malin Axelsson, Associate professor, Malmö University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MalmoU 2022
Record Dates: First submitted 2022-02-23; First posted 2022-04-04 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Fall; Pressure Ulcer; Malnutrition; Oral Health
Keywords: Prevention; Older people; Nursing care; Complex intervention
MeSH Terms: conditions — Pressure Ulcer; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Cluster randomization is going to take place via a computerized program prior to the workshops meaning that only those nurse aides, registered nurses and managers working in nursing homes allocated to the intervention group are going to develop an intervention together with the research group and then test it.
  Interventions: Behavioral: Care process for assessements of risks
- Control (No Intervention): Continue with usual care.

INTERVENTIONS:
Behavioral: Care process for assessements of risks — Intervention aiming to reduce the risk of pressure ulcers, malnutrition, poor oral health and falls among older persons in nursing homes, workshops will be conducted in collaboration with nurse aides, registered nurses and managers. Cluster randomization is going to take place via a computerized program prior to the workshops meaning that only those nurse aides, registered nurses and managers working in nursing homes allocated to the intervention group are going to develop an intervention together with the research group and then test it .
  Arms: Intervention

SUMMARY:
Inclusion criteria for study I and II is nurse aides, registered nurses and managers working in nursing homes who register in Senior Alert. To develop an intervention aiming to reduce the risk of pressure ulcers, malnutrition, poor oral health and falls among older persons in nursing homes, workshops will be conducted in collaboration with nurse aides, registered nurses and managers (study I). Cluster randomization is going to take place via a computerized program prior to the workshops meaning that only those nurse aides, registered nurses and managers working in nursing homes allocated to the intervention group are going to develop an intervention together with the research group and then test it (study II). The remaining nurse aides, registered nurses and managers working in nursing homes in the control group continue with regular care.

DETAILED DESCRIPTION:
Study I The workshops (tentative plan) Groups of one-two nurse aides, one-two registered nurses and one-two managers from the nursing homes in the intervention group will form a workshop. In total, four-five workshops will be conducted. Each workshop will begin with an introductory framing of the workshop followed by addressed activities in four stations. The activities in the four stations are designed to give the participants possibility to be active in order to develop the intervention. The participants will write down conclusions of the discussions and the discussions will be audio recorded. The written documentation and the recorded discussions will constitute data and will be analyzed using content analysis.

Station one: the participants will discuss beforehand written questions based on the results of our previous studies, and literature in order to stimulate reflection and discussion. The participants will discuss how to work in a better/different way with risk assessments, care interventions and follow-ups that can contribute to improve the preventive work so that older persons are risk assessed, get the right care interventions planned, performed and evaluated to a greater extend. They will also discuss how the organization/routines around the preventive care process be developed. The participants will write down conclusions of the discussion.

Station two: the participants will discuss beforehand written questions concerning the preventive care process according to Senior Alert. The participants will work creatively to identify barriers and challenges in the preventive care process according to Senior Alert and how this process could be done in a smoother way. The participants will write down conclusions of the discussion.

Station three: the participants will discuss how the intervention could be design. Focus of the discussion will be on the core components of the intervention, e.g. context, activity, participants, time required and implementation. The participants will write down the discussion.

Station four: summary of the workshop.

The intervention (tentative plan) The intervention will be written out in detail after the workshops have been conducted, but below is a short description in accordance with the one in the Ethical approval.

The content of the intervention will focus on the importance of prevention of the risk for pressure ulcers, malnutrition, poor oral health and falls among older persons in nursing homes and the preventive process in accordance with Senior Alert. The intervention could consist of; a work sheet to facilitate clinical decisions, new way of working, educational support, films or lectures, to meet nurse aides´, registered nurses´ and managers´ educational needs, fit into their organization and facilitate the preventive nursing care regarding these health risks.

Study II Feasibility/pilot testing the intervention The most suitable method will be applied to test and evaluate the intervention. A feasibility study could be carried out to evaluate if there are any uncertainties around the recruitment, data collection and retention or the intervention itself around the optimal content, delivery and acceptability. A pilot study could be carried out to address the main uncertainties in the development work and to indicate if further evaluation should be preceded or the intervention needs to be refined.

Evaluating the intervention To evaluate primary outcome measures, register data is going to be extracted from Senior Alert six months prior and one and six months after the intervention. Data on risk assessments and preventive interventions from the instruments available in Senior Alert (described in our previous studies) will be extracted. Additionally, background data regarding older persons in terms of biological sex, age and type of health care setting will be gathered from the registry.

Descriptive and analytic analysis will be performed in IBM SPSS Statistics Windows, Version 25 (Armonk, NY: IBM Corp) for comparisons between and within the intervention and control group.

To evaluate secondary outcome measurers all the nurse aides and registered nurses working in all the nursing homes included (both the intervention and the control group) will be invited to fill in questionnaires: the Psychosocial Aspects of Job Satisfaction questionnaire, the Perceived Stress Scale stress and the Stress of Conscience Questionnaire, at baseline (prior to the workshops) and six months after the intervention. Background data as age, gender, years of work experience and educational level will be collected. For comparisons between and within the intervention and control group before and after tests will be performed. IBM SPSS Statistics for Windows, Version 25 (Armonk, NY: IBM Corp) will be used to calculate descriptive and analytic statistics.

ELIGIBILITY:
Inclusion Criteria:

* Nursing homes registering in Senior Alert, which is a national quality registry

Exclusion Criteria:

* not meetin inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk assessments and prevention care interventions focusing on falls. | Baseline 6 months prior to intervention
  Registry data from Senior Alert based on the following assessment: Downtown Fall Risk Index.
Risk assessments and prevention care interventions focusing on pressure ulcers. | Baseline 6 months prior to intervention
  Registry data from Senior Alert based on the following assessment: The Modified Norton scale to measure risk for pressure ulcer.
Risk assessments and prevention care interventions focusing on malnutrition. | Baseline 6 months prior to intervention
  Registry data from Senior Alert based on the following assessment: The Short Form-Mini Nutritional Assessment measure malnutrition.
Risk assessments and prevention care interventions focusing on poor oral health | Baseline 6 months prior to intervention
  Registry data from Senior Alert based on the following assessment: The Revised Oral Assessment Guide (ROAG) to assess poor oral health.
Risk assessments and prevention care interventions focusing on falls. | 1 month after intervention
  Registry data from Senior Alert based on the following assessment: Downtown Fall Risk Index.
Risk assessments and prevention care interventions focusing on pressure ulcers. | 1 month after intervention
  Registry data from Senior Alert based on the following assessment: The Modified Norton scale to measure risk for pressure ulcer.
Risk assessments and prevention care interventions focusing on malnutrition. | 1 month after intervention
  Registry data from Senior Alert based on the following assessment: The Short Form-Mini Nutritional Assessment measure malnutrition.
Risk assessments and prevention care interventions focusing on poor oral health. | 1 month after intervention
  Registry data from Senior Alert based on the following assessment: The Revised Oral Assessment Guide (ROAG) to assess poor oral health.
Risk assessments and prevention care interventions focusing on falls. | 6 months after intervention
  Registry data from Senior Alert based on the following assessment: Downtown Fall Risk Index.
Risk assessments and prevention care interventions focusing on pressure ulcers. | 6 months after intervention
  Registry data from Senior Alert based on the following assessment: The Modified Norton scale to measure risk for pressure ulcer.
Risk assessments and prevention care interventions focusing on malnutrition. | 6 months after intervention
  Registry data from Senior Alert based on the following assessment: The Short Form-Mini Nutritional Assessment measure malnutrition.
Risk assessments and prevention care interventions focusing on poor oral health. | 6 months after intervention
  Registry data from Senior Alert based on the following assessment: the Revised Oral Assessment Guide (ROAG) to assess poor oral health.
Risk assessments and prevention care interventions focusing on falls. | 12 months after intervention
  Registry data from Senior Alert based on the following assessment: Downtown Fall Risk Index.
Risk assessments and prevention care interventions focusing on pressure ulcers. | 12 months after intervention
  Registry data from Senior Alert based on the following assessment: The Modified Norton scale to measure risk for pressure ulcer.
Risk assessments and prevention care interventions focusing on malnutrition. | 12 months after intervention
  Registry data from Senior Alert based on the following assessment: The Short Form-Mini Nutritional Assessment measure malnutrition.
Risk assessments and prevention care interventions focusing on poor oral health. | 12 months after intervention
  Registry data from Senior Alert based on the following assessment: The Revised Oral Assessment Guide (ROAG) to assess poor oral health.

SECONDARY OUTCOMES:
Perceived Stress Scale stress (PSS) | Baseline and six months after intervention
  Among nursing staff. 10 items scaled 0-4, higher scores indicate higher level of stress
Stress of Conscience (SCQ), | Baseline and six months after intervention
  Among nursing staff. 9 items scaled 0-5, higher scores indicate higher level of SCQ.
Psychosocial Aspects of Job Satisfaction Questionnarie | Baseline and six months after intervention
  Among nursing staff. 49 items, scaled 0-4, higher scores indicate higher level of psychosocial job satisfaction

OTHER OUTCOMES:
Feasibility test of the co-created intervention designed to reduce the evidence-base practice gap regarding prevention of the risk for pressure ulcer, malnutrition, poor oral health and falls using questionnaire data | Directly post intervention
  Data collected by a questionnaire specifically developed for evalutation of the co-created intervention called Evaluation of the intervention. The questionnaire contains 12 items on a dichtomous scale and two open questions.
Feasibility test of the co-created intervention designed to reduce the evidence-base practice gap regarding prevention of the risk for pressure ulcer, malnutrition, poor oral health and falls using interview data | Directly post intervention
  Individual and focus group interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Malin Axelsson, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neziraj M, Axelsson M, Kumlien C, Hellman P, Andersson M. The STAIR OF KNOWLEDGE-a codesigned intervention to prevent pressure ulcers, malnutrition, poor oral health and falls among older persons in nursing homes in Sweden: development of a complex intervention. BMJ Open. 2023 Aug 10;13(8):e072453. doi: 10.1136/bmjopen-2023-072453. PMID 37562934